CLINICAL TRIAL: NCT03342313
Title: Increasing in Chewing Number Reduces Energy Intake in Healthy Weight and Overweight Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Suwimol Sapwarobol, Assistant Professor, Chulalongkorn University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: Chewing and energy intake
Record Dates: First submitted 2017-11-10; First posted 2017-11-14 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Mastication

STUDY DESIGN:
Intervention Model Description: Randomized cross-over design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- healthy weight (Experimental): BMI (kg/m2) ≥ 18.5 and < 23
  Interventions: Other: Food - Sandwich
- Overweight (Experimental): BMI (kg/m2) ≥23 chewing 15 times and 50 times per bite
  Interventions: Other: Food - Sandwich

INTERVENTIONS:
Other: Food - Sandwich — Sandwich as a breakfast for testing chewing activities.

SUMMARY:
A randomized cross-over design aims to investigate chewing activities between healthy vs. overweight and determine effects chewing times on energy intake and postprandial plasma glucose and insulin. Forty-one participants were allocated into lean and overweight groups according to BMI. Phase I, Bite size (g/bite), bite rate (bites/min), chewing frequency (chews/min), and chews (chews/g food) were recorded after a sandwich breakfast. Phase II, gram of sandwich eaten ad libitum after 15 and 50 chew per bite (number from phase I) were recorded. Postprandial plasma glucose and insulin were examined at 0 (baseline), 30, 60, 90, 120 and 180 min.

DETAILED DESCRIPTION:
Forty-one eligible participants were divided into 2 groups; lean and overweight according to their BMI [lean BMI (kg/m2) ≥ 18.5 and < 23, overweight BMI ≥23]

Phase I: investigate the differences of chewing activities between healthy weight and overweight participants.

The day before the clinic visit, participants were requested to consume only portion control of fried rice with egg for their dinner at 6 -7 pm. No other foods or drinks were allowed after provided dinner. The next morning, participants arrived at the clinic between 7-8 am after a 12 hours overnight fast and a 24 hours period without exercise. Sandwich was served with 300 ml. of water for breakfast ad libitum. Foods consumed were recorded. A digital camera recorded each participants chewing activities including bite size (g/bite); the ratio of food weight to bite number, bite rate (bites/min); the ratio of bite number to meal time, chewing frequency (chews/min); the ratio of chews to meal time, chews (chews/g food); the ratio of chews to meal weight.

Phase II: investigate the effects 15 chews and 50 chews on energy intake, hunger, satiety, appetite, postprandial plasma glucose and insulin in both healthy weight and overweight participants Participants were allocated into 2 groups of a 15 chews and 50 chews per bites with 2 weeks of wash-out period. The day before the clinic visit, participants were requested to consume only portion control of fried rice with egg for their dinner at 6 -7 pm. No other foods or drinks were allowed after provided dinner in order to prevent confounding factors of previous food consumption. On the next day, participants arrived at the clinic between 7-8 am after a 12 hours overnight fast and a 24 hours period without exercise. At clinic visit, baseline characteristics including anthropometry, hunger, satiety, appetite, and plasma glucose and insulin concentrations were collected before breakfast was served. Participant was requested to rate their hunger, satiety and appetite using a visual analogue scale (VAS) questionnaire.

After collecting baseline indicators, participants were served an ad libitum sandwich and 300 ml water for breakfast. Participants had to finish their breakfast within 20 min after first bite. VAS questionnaire and blood samples of postprandial glucose and insulin were examined at 0 (baseline) 30, 60, 90, 120 and 180 min after test meal. Blood samples was collected from indwelling catheters at mentioned time points.

ELIGIBILITY:
Inclusion Criteria:

* non-smoking
* eating breakfast regularly
* not allergic to any food
* no eating disorders
* weight stable over the past 3 months

Exclusion Criteria:

* have dental problem
* taking any medications or dietary supplements that may confound any study indicators

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2015-03-15 (Actual); Primary Completion 2015-08-18 (Actual); Study Completion 2016-02-04 (Actual)

PRIMARY OUTCOMES:
chewing times per bite | 2 months
  chewing times per bite

SECONDARY OUTCOMES:
energy intake | 2 months
  chewing 15 and 50 times per bite on amount of food eaten
hunger, satiety, appetite | 2 months
  a paper- based visual analogue scale (VAS) questionnaire of hunger, satiety, appetite. Each VAS questionnaire contains 100 millimeters in length and labels from not at all (scores 0) to extremely (scores10).
postprandial plasma glucose | at 0, 30, 60, 90, 120 and 180 min after eating
  blood glucose after eating
postprandial plasma insulin | at 0, 30, 60, 90, 120 and 180 min after eating
  plasma insulin after eating

CONTACTS AND LOCATIONS:
Overall Officials: suwimol sapwarobol, Principal Investigator — Chulalongkorn University
Locations (1):
- Suwimol Sapwarobol, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li J, Zhang N, Hu L, Li Z, Li R, Li C, Wang S. Improvement in chewing activity reduces energy intake in one meal and modulates plasma gut hormone concentrations in obese and lean young Chinese men. Am J Clin Nutr. 2011 Sep;94(3):709-16. doi: 10.3945/ajcn.111.015164. Epub 2011 Jul 20. PMID 21775556